CLINICAL TRIAL: NCT01356849
Title: RADAR: Reducing Residual Albuminuria in Subjects With Diabetes and Nephropathy With AtRasentan - A Phase 2b, Prospective, Randomized, Double-Blind, Placebo-Controlled Trial to Evaluate Safety and Efficacy
Brief Title: Evaluate the Efficacy and Safety of Once Daily Administration of Atrasentan Tablets (Low and High) Compared to Placebo in Reducing Residual Albuminuria in Type 2 Diabetic Patients With Nephropathy Who Are Treated With the Maximum Tolerated Labeled Dose of a Renin Angiotensin System (RAS) Inhibitor
Acronym: RADAR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M11-350
Record Dates: First submitted 2011-04-19; First posted 2011-05-20 (Estimated); Last update posted 2013-08-28 (Estimated); Status verified 2013-08

CONDITIONS: Chronic Kidney Disease; Diabetic Nephropathy
Keywords: Endothelin Receptor Antagonists; Proteinuria
MeSH Terms: conditions — Renal Insufficiency, Chronic; Diabetic Nephropathies; Proteinuria | interventions — Atrasentan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group A - Placebo QD (Placebo Comparator)
  Interventions: Drug: Placebo
- Group B - Low dose Atrasentan QD (Active Comparator)
  Interventions: Drug: Atrasentan
- Group C - High dose Atrasentan QD (Active Comparator)
  Interventions: Drug: Atrasentan

INTERVENTIONS:
Drug: Atrasentan — Subjects will take two tablets daily of either low dose Atrasentan QD or high dose Atrasentan QD for 12 weeks during the treatment period.
  Other Names: ABT-627
  Arms: Group B - Low dose Atrasentan QD; Group C - High dose Atrasentan QD
Drug: Placebo — Subjects will take two tablets daily of placebo QD for 12 weeks during the treatment period.
  Arms: Group A - Placebo QD

SUMMARY:
Prospective, Randomized, Double-Blind, Placebo-Controlled Multicenter Study. The objective of the study is to evaluate the efficacy and safety of once daily administration of atrasentan tablets (low dose and high dose) compared to placebo in reducing residual albuminuria in Type 2 diabetic patients with nephropathy who are treated with the maximum tolerated labeled dose of a Renin Angiotensin System (RAS) inhibitor. If the patient is already receiving a maximum tolerated labeled daily dose of RAS inhibitor and a diuretic, he/she will complete 4 weeks of the Run-in Period on a dose that has not been adjusted. If the patient is currently not receiving a maximum labeled daily dose of a RAS inhibitor then the dose will be titrated up to the maximum tolerated labeled dose over the course of 4 to 8 weeks during the Run-in Period. It is expected that subjects not receiving a diuretic will have a diuretic added or titrated during this period to maximize RAS inhibition. Following titration to the maximum tolerated labeled dose, the patient will complete an additional 4 weeks of Run-In Period on an unchanged doses of RAS inhibitor and diuretics, unless medically contraindicated. The randomization will be stratified based on country where subjects are enrolled into the study, and the Week -1 Urinary Albumin to Creatinine Ratio (UACR) levels (< or = 1000 mg/g [113 mg/mmol], or > 1000 mg/g [113 mg/mmol]). Within each stratum, subjects will be randomly assigned in a 1:2:2 ratio to one of the following blinded treatment groups: Group A - Placebo once daily (QD) Group B - low dose atrasentan QD Group C - high dose atrasentan QD After the 12 weeks of study drug treatment, subjects will be followed up to 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patient is > or = 18 years old.
* Patient has Type 2 diabetes and has been treated with at least one anti hyperglycemic medication within the 12 months prior to the Screening Period.
* Patient is currently receiving an angiotensin converting enzyme inhibitor (ACEi) or Angiotensin II receptor blocker (ARB) (Renin Angiotensin System (RAS) inhibitor).
* For entry in the Run-in Period the patient must satisfy the following criteria based on the Screening laboratory values:

  * Estimated glomerular filtration rate (eGFR) ≥ 30 and ≤ 75 mL/min/1.73m2 by Epidemiology Collaboration (EPI) formula
  * Urinary Albumin to Creatinine Ratio (UACR) > or = 300 and < or = 3500 mg/g as determined by the geometric mean of the two morning void urine specimens obtained at the Screening visit (UACR > or = 34 mg/mmol and < or = 396 mg/mmol)
  * Serum albumin > or = 3.0 g/dL (30 g/L) - B-type Natriuretic Peptide (BNP) < or = 200 pg/mL (57.8 pmol/L) * Negative serum pregnancy test for female patients
  * Systolic Blood Pressure (SBP) > or = 110 mmHg and < or = 180 mmHg
  * Glucosylated hemoglobin A1c (HbA1c) < or = 12%
* For entry in the Treatment Period the patient must satisfy the following criteria based on the last visit of the Run-in Period laboratory values:

  * Renin Angiotensin System (RAS) inhibitor at maximum tolerated labeled dose for the previous 4 weeks with no adjustments of dose
  * Diuretic at any dose unless medically contraindicated (with the exception of loop diuretics > or = 120 mg QD of furosemide or > or = 3.0 mg QD of bumetanide or > or = 150 mg QD of ethacrynic acid or > or = 60 mg QD of torasemide)
  * Urinary Albumin to Creatinine Ratio (UACR) > or = 200 and < or = 3500 mg/g as determined by the median of the three morning void urine specimens obtained prior to the Week -1 visit (UACR > or = 23 mg/mmol and < or = 396 mg/mmol)
  * Systolic blood pressure (SBP) > or = 110 mmHg and < or = 160 mmHg
  * Serum Potassium < or = 5.5 mEq/L (5.5 mmol/L)
  * Negative serum pregnancy test for female patients

Exclusion Criteria:

* Patient has a history of moderate or severe edema, facial edema unrelated to trauma, or a history of myxedema in the prior 6 months to Screening.
* Patient is receiving loop diuretics > or = 120 mg QD of furosemide or > or = 3.0 mg QD of bumetanide or > or = 150 mg QD of ethacrynic acid or > or = 60 mg QD of torasemide.
* Patient has a history of pulmonary edema.
* Patient has a history of pulmonary hypertension, or any lung diseases requiring oxygen therapy (i.e., chronic obstructive pulmonary disease, emphysema, pulmonary fibrosis).
* Patient has a history of orthostatic hypotension within the past 6 months as defined by the presence of a supine-to-standing blood pressure decrease > or = 20 mmHg systolic or > or = 10 mmHg diastolic within 3 minutes of standing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2011-04; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline to Week 12 in Urinary Albumin to Creatinine Ratio (UACR) | Every two weeks for 12 weeks

SECONDARY OUTCOMES:
Differences in change from baseline to each post baseline measure for estimated glomerular filtration rate (eGFR) | Every two weeks for 12 weeks
Differences in change from baseline to each post baseline measure for EQ-5D Index Score | Once a month for 3 months
Differences in change from baseline to each post baseline measure for each of the Kidney Disease Quality of Life (KDQOL) Kidney Disease Targeted Scales | Once a month for 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Blai Coll, MD, Study Director — AbbVie
Locations (72):
- United States (59):
  - Site Reference ID/Investigator# 46345, Pell City, Alabama
  - Site Reference ID/Investigator# 46035, Tempe, Arizona
  - Site Reference ID/Investigator# 46016, Azusa, California
  - Site Reference ID/Investigator# 45992, Chula Vista, California
  - Site Reference ID/Investigator# 46000, La Mesa, California
  - Site Reference ID/Investigator# 46038, Lincoln, California
  - Site Reference ID/Investigator# 45994, Long Beach, California
  - Site Reference ID/Investigator# 45998, Los Angeles, California
  - Site Reference ID/Investigator# 47584, Los Gatos, California
  - Site Reference ID/Investigator# 64465, National City, California
  - Site Reference ID/Investigator# 65862, Orange, California
  - Site Reference ID/Investigator# 46019, Riverside, California
  - Site Reference ID/Investigator# 46110, Salinas, California
  - Site Reference ID/Investigator# 46017, Yuba City, California
  - Site Reference ID/Investigator# 46662, Westminster, Colorado
  - Site Reference ID/Investigator# 46033, Coral Gables, Florida
  - Site Reference ID/Investigator# 45989, Hialeah, Florida
  - Site Reference ID/Investigator# 46667, Lauderdale Lakes, Florida
  - Site Reference ID/Investigator# 46123, Miami, Florida
  - Site Reference ID/Investigator# 46115, Ocala, Florida
  - Site Reference ID/Investigator# 46664, Pembroke Pines, Florida
  - Site Reference ID/Investigator# 46031, Pembroke Pines, Florida
  - Site Reference ID/Investigator# 46040, Pembroke Pines, Florida
  - Site Reference ID/Investigator# 46122, Port Charlotte, Florida
  - Site Reference ID/Investigator# 46015, West Palm Beach, Florida
  - Site Reference ID/Investigator# 50482, Jonesboro, Georgia
  - Site Reference ID/Investigator# 46034, Meridian, Idaho
  - Site Reference ID/Investigator# 46666, Chicago, Illinois
  - Site Reference ID/Investigator# 45996, Evergreen Park, Illinois
  - Site Reference ID/Investigator# 46002, Gurnee, Illinois
  - Site Reference ID/Investigator# 46111, Shreveport, Louisiana
  - Site Reference ID/Investigator# 46030, Oxon Hill, Maryland
  - Site Reference ID/Investigator# 45991, Rockville, Maryland
  - Site Reference ID/Investigator# 46025, Novi, Michigan
  - Site Reference ID/Investigator# 46023, Brooklyn Center, Minnesota
  - Site Reference ID/Investigator# 46062, Farmington, Missouri
  - Site Reference ID/Investigator# 48942, Omaha, Nebraska
  - Site Reference ID/Investigator# 46349, Omaha, Nebraska
  - Site Reference ID/Investigator# 46116, Las Vegas, Nevada
  - Site Reference ID/Investigator# 50483, Albany, New York
  - Site Reference ID/Investigator# 68328, New Hyde Park, New York
  - Site Reference ID/Investigator# 65863, Asheville, North Carolina
  - Site Reference ID/Investigator# 50529, Greensboro, North Carolina
  - Site Reference ID/Investigator# 46129, Greenville, North Carolina
  - Site Reference ID/Investigator# 46022, Morehead City, North Carolina
  - Site Reference ID/Investigator# 46224, Doylestown, Pennsylvania
  - Site Reference ID/Investigator# 46028, Orangeburg, South Carolina
  - Site Reference ID/Investigator# 46702, Orangeburg, South Carolina
  - Site Reference ID/Investigator# 46024, Greenville, Texas
  - Site Reference ID/Investigator# 46228, Houston, Texas
  - Site Reference ID/Investigator# 47068, Houston, Texas
  - Site Reference ID/Investigator# 64464, Houston, Texas
  - Site Reference ID/Investigator# 64483, Mission, Texas
  - Site Reference ID/Investigator# 46348, San Antonio, Texas
  - Site Reference ID/Investigator# 46063, San Antonio, Texas
  - Site Reference ID/Investigator# 68486, San Antonio, Texas
  - Site Reference ID/Investigator# 46669, Bennington, Vermont
  - Site Reference ID/Investigator# 46026, Alexandria, Virginia
  - Site Reference ID/Investigator# 46027, Fairfax, Virginia
- Canada (3):
  - Site Reference ID/Investigator# 67762, Kitchener
  - Site Reference ID/Investigator# 50526, Sarnia
  - Site Reference ID/Investigator# 50525, Thornhill
- Puerto Rico (8):
  - Site Reference ID/Investigator# 47067, Caguas
  - Site Reference ID/Investigator# 50522, Manatí
  - Site Reference ID/Investigator# 46352, Ponce
  - Site Reference ID/Investigator# 46351, Ponce
  - Site Reference ID/Investigator# 46133, Ponce
  - Site Reference ID/Investigator# 46131, Rio Piedras
  - Site Reference ID/Investigator# 46132, San Juan
  - Site Reference ID/Investigator# 46230, Santurce
- Taiwan (2):
  - Site Reference ID/Investigator# 51566, Taichung
  - Site Reference ID/Investigator# 51567, Taichung

REFERENCES:
- [Derived] Smeijer JD, Kohan DE, Rossing P, Correa-Rotter R, Liew A, Tang SCW, de Zeeuw D, Gansevoort RT, Ju W, Lambers Heerspink HJ. Insulin resistance, kidney outcomes and effects of the endothelin receptor antagonist atrasentan in patients with type 2 diabetes and chronic kidney disease. Cardiovasc Diabetol. 2023 Sep 16;22(1):251. doi: 10.1186/s12933-023-01964-8. PMID 37716952
- [Derived] Lin CW, Mostafa NM, L Andress D, J Brennan J, Klein CE, Awni WM. Relationship Between Atrasentan Concentrations and Urinary Albumin to Creatinine Ratio in Western and Japanese Patients With Diabetic Nephropathy. Clin Ther. 2018 Feb;40(2):242-251. doi: 10.1016/j.clinthera.2017.07.011. Epub 2017 Jul 27. PMID 28756065